CLINICAL TRIAL: NCT05125913
Title: Long Term Cardio-Vascular Risk Assessment in CKD and Kidney Transplanted Patients Following SARS-COV-2 Disease: CARDIO SCARS IN CKD Protocol for a Multi-center Observational Match Controlled Trial
Brief Title: Long Term Cardio-Vascular Risk Assessment in CKD and Kidney Transplanted Patients Following SARS-COV-2
Acronym: CARDIO SCARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, Principal Investigator, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: Cardio Scars
Record Dates: First submitted 2021-11-10; First posted 2021-11-18 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: CKD; Dialysis; Kidney Transplant; COVID-19; Cardiovascular Disease; Endothelial Dysfunction
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases | interventions — Vascular Stiffness; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 group: Patients with CKD stage 3-5, on dialysis or kidney transplanted patients with confirmed SARS-CoV-2 infection by reverse transcriptase polymerase chain reaction (RT-PCR), at minimum 2 weeks after the confirmed test.
  Interventions: Diagnostic Test: FMD; Diagnostic Test: Arterial stiffness; Diagnostic Test: Assessment of IMT; Diagnostic Test: Echocardiography; Diagnostic Test: LUS; Diagnostic Test: BIS analysis; Other: Biomarkers determination
- non-COVID-19 group: CKD stage 3-5, dialysis or kidney transplantation matched patients without confirmed SARS-CoV-2 infection
  Interventions: Diagnostic Test: FMD; Diagnostic Test: Arterial stiffness; Diagnostic Test: Assessment of IMT; Diagnostic Test: Echocardiography; Diagnostic Test: LUS; Diagnostic Test: BIS analysis; Other: Biomarkers determination

INTERVENTIONS:
Diagnostic Test: FMD — Measurements will be made by using ultrasound system with a 12-Mhz probe. All vasoactive medications will be withheld for 24 h before the procedure. The participants will remain at rest in the supine position for at least 15 minutes before the examination. Each subject's right arm will be comfortably immobilized in the extended position to allow consistent recording of the brachial artery 2-4 cm above the antecubital fossa. If an arteriovenous fistula is present, the contralateral arm will be used for assessment. Three adjacent measurements of end-diastolic brachial artery diameter will be made from single 2D frames. The maximum FMD diameters will be calculated as the average of the three consecutive maximum diameter measurements after hyperemia and nitroglycerin, respectively.
Diagnostic Test: Arterial stiffness — Arterial stiffness assessment will be performed by applanation tonometry with the patient being recumbent, 10 minutes before the measures were done. The carotid and femoral pulse will be acquired by applanation tonometry sequentially, allowing a single operator to acquire the measurement. The transit time from the R-wave of the simultaneously acquired electrocardiogram to the foot of the carotid and femoral pulse is measured. The difference-acquired electrocardiogram to the foot of the carotid and femoral pulse is measured. The difference between these 2 transit times is divided by distances measured from the body surface to estimate the arterial path length in order to calculate carotid-femoral PWV.
Diagnostic Test: Assessment of IMT — A high-resolution B-mode ultrasound of the common carotid arteries with scanning of the longitudinal axis until the bifurcation and of the transversal axis will be performed using ultrasonic pulse with a middle frequency of 12 MHz. For each carotid artery, two longitudinal measurements will be obtained by rotating the vessels at 180o increments along their axis. IMT will be measured at 1 cm proximal to the bifurcation on each side.
Diagnostic Test: Echocardiography — Echocardiography will be performed on each patient at baseline; the measurements will be carried out according to the recommendations of the American Society of Echocardiography by an observer unaware of the lung ultrasound and bioimpedance results. Echocardiographic evaluation will provide information about cardiac anatomy (e.g. volumes, geometry, mass) and function (e.g. left ventricular function and wall motion, valvular function, right ventricular function, pulmonary artery pressure, pericardium).
Diagnostic Test: LUS — Examinations will be performed in the supine position. Scanning of the anterior and lateral chest will be performed on both sides of the chest, from the second to the fourth (on the right side to the fifth) intercostal spaces, at parasternal to mid-axillary lines. B-lines will be recorded in each intercostal space and were defined as a hyperechoic, coherent US bundle at narrow basis going from the transducer to the limit of the screen. B-lines starting from the pleural line can be either localized or scattered to the whole lung and be present as isolated or multiple artifacts. The sum of B-lines produces a score reflecting the extent of lung water accumulation (0 being no detectable B-line).
Diagnostic Test: BIS analysis — This analysis will be performed at baseline using the portable whole-body multifrequency bioimpedance analysis device using specific electrodes. Based on a fluid model using 50 discrete frequencies (5-1000kHz), the extracellular water (ECW), the intracellular water (ICW) and the total body water (TBW) are calculated. These volumes are then used to determine the amount of fluid overload. All calculations are automatically performed by the software of the BCM® device. Absolute fluid overload (AFO) is defined as the difference between the expected patient's ECW under normal physiological conditions and the actual ECW, whereas the relative fluid overload (RFO) is defined as the absolute fluid overload AFO to ECW ratio.
Other: Biomarkers determination — Biomarkers by ELISA: IL-1, IL-6, VCAM1, Endoglin, NO and ADMA

SUMMARY:
The occurrence of novel coronavirus disease 2019 (COVID-19), caused by the Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2), has offered an unmatched global challenge for the healthcare research community. SARS-CoV-2 infection is produced by binding to angiotensin-converting enzyme (ACE2), which among other sites is highly expressed in the endothelial cells of the blood vessels, pericytes and the heart, as well as in renal podocytes and proximal tubular epithelial cells. Autopsy studies detected the presence of SARS-CoV-2 in both myocardium and renal tissue, suggesting that COVID-19 profoundly influences the cardiovascular (CV) system and the kidneys and this may lead to long-termed cardio-pulmonary-renal consequences. Data emerging from the general population suggests that COVID-19 is essentially an endothelial disease, with possible deleterious long-term effects that are currently incompletely understood. Therefore, the investigators aim to assess the CV risk in a chronic kidney disease (CKD) including dialysis patients and kidney transplanted (KTx) population, following SARS-CoV-2 infection, by determining the long-term impact of this disease on CV and renal outcomes in the aforementioned population as compared to a control group of matched patients.

DETAILED DESCRIPTION:
The coronavirus disease caused by the SARS-CoV-2 first emerged in early December 2019 and was declared a pandemic on March 2020. SARS-CoV-2 infection is produced by binding to ACE2, which among other sites is highly expressed in the endothelial cells of the blood vessels, pericytes and the heart, as well as in renal podocytes and proximal tubular epithelial cells. Of note, ACE2 RNA expression in kidney is nearly 100-fold higher than that in lungs. COVID-19 and cardiovascular disease (CVD) seem to be interconnected; on the one hand, prior CVD as well as CV risk factors are associated with an increased incidence of the disease (with fatal outcomes) and on the other hand COVID-19 can exacerbate associated CVD and determine de novo cardiac complications (acute myocardial injury, stress cardiomyopathy, myocarditis, pericarditis, arrhythmias, heart failure and cardiogenic shock). At the same time, COVID-19 disease can lead to acute kidney injury directly, or due to sepsis, multi-organ failure and shock. The preexistence of both CVD and CKD is associated with a higher risk of severe disease and worse prognosis. CKD patients are already at high risk for CV complications with CVD the leading cause of morbidity and mortality in CKD.

The reported incidence of thrombotic complications in patients with COVID-19 varies between studies, ranging from 25% to 42.6%. It is still under debate if these hemostatic changes are a particular effect of SARS-CoV-2, the inflammatory response, or if they appear secondary to either endothelial dysfunction (ED) or sepsis. Prolonged hypoxemia, cytokine storm and local pulmonary thrombotic phenomena, as well as the associated liver dysfunction secondary to the viral binding to a hepatic receptor are some of the COVID-19's peculiarities that can lead to a higher thrombotic burden. Infection of endothelial cells or perycites is of particular importance because this could lead to severe microvascular and macrovascular dysfunction. ED refers to a systemic condition in which the endothelium loses its physiological properties, including the tendency to promote vasodilation, fibrinolysis, and anti-aggregation. Morphologic findings from deceased patients confirm the presence of viral elements within endothelial cells and an accumulation of inflammatory cells, with evidence of endothelial and inflammatory cell death. Endothelitis in several organs as a direct consequence of viral involvement and of the host inflammatory response may explain the impaired microcirculatory function in different vascular beds and clinical sequel in patients with COVID-19.

The COVID-19 pandemic is forcing healthcare systems and societies to scrutinize how care is delivered and valuable lessons are being learned. Furthermore, as mentioned above, the assessment of CV risk is crucially important for these patients. In this regard, a bedside assembly of reliable and thorough investigations that will provide lasting insights past the time of this pandemic, can become a very valuable tool.

The overall scope of this study is to assess the CV risk in a CKD (stage 3 to 5D) and kidney transplanted population, following COVID-19 infection, with focus on the ED as compared to a control group of matched patients. By using clinical evaluation, flow-mediated dilatation (FMD), pulse wave velocity (PWV), intima media thickness (IMT), echocardiographic parameters, Lung ultrasonography (LUS), bioimpedance spectroscopy (BIS) derived fluid status parameters (over hydration, total body water, extracellular water and intracellular water) and a series of novel biomarkers, the investigators intent to determine the long-term impact of this disease on CV and renal outcomes in the aforementioned population.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years;
* Patients with CKD stage 3-5, patients on dialysis or KTx patients with confirmed COVID-19, at minimum 2 weeks after the confirmed test;
* Age, sex and kidney disease (CKD stage 3-5, dialysis or KTx) matched patients without confirmed SARS-CoV-2 infection.

Exclusion Criteria:

* Prior diagnosis of pulmonary fibrosis, pneumectomy or massive pleural effusion;
* Active malignancies.
* Pregnancy;
* Active systemic infections (due to difficulties in the interpretation of nonspecific inflammation biomarkers in this type of patients);
* Congenital heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective case-control study will include CKD stage 3 to 5 patients, dialysis patients and KTx patients.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 24 months post-COVID-19
  One of the primary outcome of this study will be all-cause mortality rate.
MACE | 24 months post-COVID-19
  Another primary outcome will be a composite CV outcome (time to first non-fatal myocardial infarction, non-fatal stroke, and hospitalization for heart failure or CV death).
Endothelial dysfunction | 6 months post-COVID-19
  The investigators will determine long-term impact of the COVID-19 on markers of CV risk and ED in all included patients.
Endothelial dysfunction | 12 months post-COVID-19
  The investigators will determine long-term impact of the COVID-19 on markers of CV risk and ED in all included patients.
Endothelial dysfunction | 24 months post-COVID-19
  The investigators will determine long-term impact of the COVID-19 on markers of CV risk and ED in all included patients.

SECONDARY OUTCOMES:
Renal outcome | 6 months post-COVID-19
  Secondary outcomes are defined as a composite of renal outcome: doubling of creatinine or a 40% decline in eGFR or dialysis initiation in CKD or KTx patients.
Renal outcome | 12 months post-COVID-19
  Secondary outcomes are defined as a composite of renal outcome: doubling of creatinine or a 40% decline in eGFR or dialysis initiation in CKD or KTx patients.
Renal outcome | 24 months post-COVID-19
  Secondary outcomes are defined as a composite of renal outcome: doubling of creatinine or a 40% decline in eGFR or dialysis initiation in CKD or KTx patients.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian C Covic, Professor, Study Director — Grigore T. Popa University of Medicine and Pharmacy
Locations (1):
- Dr CI Parhon Clinical Hospital of Iasi, Iași, Romania

REFERENCES:
- [Derived] Tapoi L, Apetrii M, Dodi G, Nistor I, Voroneanu L, Siriteanu L, Onofriescu M, Kanbay M, Covic A. Long-term cardio-vascular risk assessment in chronic kidney disease and kidney transplanted patients following SARS-COV-2 disease: protocol for multi-center observational match controlled trial. BMC Nephrol. 2022 May 6;23(1):176. doi: 10.1186/s12882-022-02809-4. PMID 35524223